CLINICAL TRIAL: NCT02410876
Title: Changes of microRNA Expression in Obstructive and Neurogenic Bladder Dysfunction Reveal Common Signalling Pathways Relevant for Disease Progression and Recovery
Brief Title: Changes of microRNA Expression in Obstructive and Neurogenic Bladder Dysfunction
Acronym: MoVe
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Swiss National Science Foundation (Other); Balgrist University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 331/2014
Record Dates: First submitted 2015-04-02; First posted 2015-04-08 (Estimated); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Disorder of the Lower Urinary Tract
Keywords: Bladder; neurogenic lower urinary tract dysfunction; benign prostatic obstruction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — cold cup biopsies of the bladder wall
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Controls: No lower urinary tract symptoms undergoing cystoscopy in anesthesia for stone treatment or microhematuria assessment.
  Interventions: Procedure: Bladder biopsy
- Spinal cord injury/acontractile: Patients with traumatic spinal cord injury (SCI) with no (neither spontaneous nor provoked) detrusor activity during the filling phase of urodynamics.
  Bladder biopsy 6 weeks after trauma 6 months later urodynamic study and bladder biopsy
  Interventions: Procedure: Bladder biopsy; Procedure: Urodynamic study
- Spinal cord injury/Detrusor overactivity: SCI patients with proven detrusor (urodynamics) overactivity during the filling phase.
  Bladder biopsy 6 weeks after trauma 6 months later urodynamic study and bladder biopsy
  Interventions: Procedure: Bladder biopsy; Procedure: Urodynamic study
- Prostatic obstruction/acontractile: Low flow to no flow, no measurable detrusor activity on urodynamic evaluation, cystoscopy in line with obstruction.
  Bladder biopsy at TURP (transurethral resection prostate) 3 months later urodynamic study and bladder biopsy
  Interventions: Procedure: Bladder biopsy; Procedure: Urodynamic study
- Prostatic obstruction/ obstructed: Obstruction according to Schäfer nomogram on urodynamic evaluation. Bladder biopsy at TURP 3 months later urodynamic study and bladder biopsy
  Interventions: Procedure: Bladder biopsy; Procedure: Urodynamic study

INTERVENTIONS:
Procedure: Bladder biopsy — Small biopsy of the bladder is taken with cold-cup tongs.
Procedure: Urodynamic study — Assessment of bladder function through intravesical and intrabdominal pressure measurements according to International Continence Society standards.
  Groups: Prostatic obstruction/ obstructed; Prostatic obstruction/acontractile; Spinal cord injury/Detrusor overactivity; Spinal cord injury/acontractile

SUMMARY:
Patients with obstructive or neurogenic lower urinary tract disease will be invited to participate. Upon agreement they will undergo an assessment of bladder function (questionnaires) and bladder biopsies at 2 time-points. Bladder biopsies will be evaluated for molecular changes in the laboratory and compared to the functional findings.By uncovering the molecular similarities and differences between BLUTD and NLUTD, the investigators will elucidate some of the causative factors in the development of these disorders and highlight the impact of myogenic and neurogenic components postulated to be involved. The project involves close collaboration between clinical and basic research.

DETAILED DESCRIPTION:
Lower urinary tract dysfunction (LUTD) has multiple causes including bladder outlet obstruction (BOO) as a result of benign prostatic hyperplasia (BPH) and neurological diseases including spinal cord injury (SCI). Manifestations of LUTD include storage symptoms such as increased daytime frequency, nocturia, urgency and urinary incontinence and voiding symptoms such as slow stream, hesitancy and incomplete emptying. The consequences of both BOO-induced (BLUTD) and neurogenic LUTD (NLUTD), leading to functional entities including the low compliance high pressure bladder as well as the acontractile high volume low pressure bladder, are believed to share some pathogenetic mechanisms.

In a previous project, the investigators have established micro ribonucleic acid (miRNA) and messenger ribonucleic acid (mRNA) expression profiles of several urodynamically defined states of BLUTD. In this follow-up project, the investigators propose to extend these studies, undertaking a comparative miRNA and RNA profiling of BLUTD and NLUTD, and investigate the dynamic alteration of microRNA expression in different functional manifestations of disease. The investigators propose to validate primary gene targets of miRNAs differentially expressed in urodynamically defined states of BLUTD and identify signaling pathways, activated during the progression from hypertrophy to decompensation. Monitoring the reversal of changes in miRNA expression after relief of obstruction and restoration of normal bladder function will help delineate the key BOO-induced miRNAs with regulatory potential. Similarly, the dynamics of miRNA alteration, observed in SCI patients during the development and management of NLUTD should reveal the role of miRNA in gene expression regulation during neurogenic-induced organ remodelling.

By uncovering the molecular similarities and differences between BLUTD and NLUTD, the investigators will elucidate some of the causative factors in the development of these disorders and highlight the impact of myogenic and neurogenic components postulated to be involved. The project involves close collaboration between clinical and basic research, and combines the analysis of human biopsy material with in vitro cell-based assays, creating a comprehensive platform for the dissection of molecular mechanisms of LUTD. This project will keep the momentum of the investigators' previous research and contribute to the basic and applied studies into bladder remodeling. It is a logical continuation of their on-going studies of the role of miRNAs in LUT disorders but represents a novel direction of research and has high diagnostic and therapeutic potential.

ELIGIBILITY:
Inclusion Criteria:

* Planned cystoscopy in anesthesia for upper tract stone treatment or microscopic hematuria evaluation (controls)
* Planned TURP (transurethral prostate resection) (BLUTD)
* Spinal cord injury (in last 6 weeks) (NLUTD)
* Prior urodynamic study
* Informed consent

Exclusion Criteria:

* Age < 18 years old
* Pregnancy
* Urinary tract infection
* History of or current genitourinary tuberculosis, bladder malignancy, radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Controls: patients with cystoscopy for stone disease or microhematuria without bladder symptoms Patients with spinal cord injury or benign prostatic obstruction.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-06; Primary Completion 2020-12 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Establishment of mRNA targets and pathways defining a disease state and/or potentially amendable to pharmacological evaluation. | 8 years
  Next generation sequencing of bladder wall tissue to determine changes in mRNAs and their targets and pathways

CONTACTS AND LOCATIONS:
Overall Officials: Fiona C Burkhard, MD, Principal Investigator — Insel Gruppe AG, University Hospital Bern; Jürgen Pannek, MD, Principal Investigator — Swiss paraplegic center Nottwil
Locations (1):
- University Hospital Inselspital, Bern, Switzerland